CLINICAL TRIAL: NCT00002321
Title: A Phase I Study of the Safety of Proleukin (Aldesleukin) in Combination With Ganciclovir and Antiretroviral Therapy in HIV Seropositive Patients With Cytomegalovirus (CMV) Retinitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 086A; CS-L293-10
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Interleukin-2; Ganciclovir; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
To determine the MTD and dose-limiting toxicities of a regimen of therapeutic ganciclovir, antiretroviral therapy, and recombinant interleukin-2 (aldesleukin; Proleukin) as an immune adjuvant in HIV-seropositive patients. To investigate the effect of increasing doses of Proleukin on the time to progression of CMV retinitis in patients being treated with therapeutic ganciclovir and antiretroviral therapy. To evaluate the incidence and level of anti-IL-2 antibody formation to subcutaneously administered Proleukin in this patient population.

DETAILED DESCRIPTION:
Patients will receive subcutaneous Proleukin in combination with ganciclovir and antiretroviral therapy, and the MTD will be determined.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

Documented HIV seropositivity.

Prior Medication:

Required:

* FDA-approved antiretroviral therapy for at least 2 months prior to study entry.

Allowed:

* Prior G-CSF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Med College of Ohio, Toledo, Ohio, United States